CLINICAL TRIAL: NCT03864757
Title: APrevent Vocal Implant System (VOIS) for Adjustable Treatment of Unilateral Vocal Fold Paralysis (UVFP) - an Open-label, Non-randomized Pilot Study
Brief Title: APrevent Vocal Implant System (VOIS) for Adjustable Treatment of Unilateral Vocal Fold Paralysis (UVFP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: APrevent Biotech GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: APrevent-VOIS-Implant-001
Record Dates: First submitted 2019-02-26; First posted 2019-03-06 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Paralysis, Unilateral, Vocal Cord
Keywords: unilateral vocal fold paralysis; type I thyroplasty
MeSH Terms: conditions — Vocal Cord Paralysis | interventions — Laryngoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UVFP correction surgery (Experimental): Short-term implantation of VOIS and evaluation of voice quality and glottal closure.
  Interventions: Device: thyroplasty implant

INTERVENTIONS:
Device: thyroplasty implant — Short-term implantation of thyroplasty implant, VOIS, and evaluation of voice quality and glottal closure. After evaluation, remove VOIS and perform medialization of vocal folds using conventional thyroplasty.

SUMMARY:
The objective of this study is to evaluate pre- and intraoperative voice quality, the degree of vocal fold closure and the Maximum Phonation Time (MPT), first determined after temporary APrevent® VOIS implantation and then after permanent existing product implantation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18 and 80 years
* Diagnosed with permanent UVFP and insufficient glottal closure and planned type I thyroplasty with conventional implant
* Ability to co-operate with the investigator and to comply with the requirements of the entire study

Exclusion Criteria:

* Any other significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the clinical investigation may influence the result of the clinical investigation, or the participant's ability to participate in the clinical investigation
* Scheduled elective surgery or other procedures requiring general anaesthesia during clinical investigation
* Had medialization thyroplasty before
* Had injection medialization laryngoplasty in the past two years.
* Presence of structural vocal fold lesions such as polyp or nodules
* Status post total cordectomy
* Previous laryngeal framework surgery (any type of thyroplasty, arytenoid adduction)
* Significant non-laryngeal speech abnormality (severe dysarthria determined by a panel of trained speech therapists)
* Severe coagulopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
Change in voice quality by RBH-Scale | pre-surgery, right after temporarily implantation
  Roughness(R), Breathiness(B), Hoarseness(H) Scale will be rated on a 4-point severity scale (0, normal; 1, mild deviance; 2, moderate deviance; and 3, severe deviance).
Change in Glottal closure by Södersten and Lindestad classification | pre-surgery, right after temporarily implantation
Change in maximum phonation time in seconds | pre-surgery, right after temporarily implantation
  The prolongation of a/a:/, for as long as possible after maximal inspiration, and at a spontaneous, comfortable pitch and loudness.

SECONDARY OUTCOMES:
Evaluation of surgical handling and device fitting using a VAS scale | right after temporarily implantation
  Visual analogue scale(VAS) of Subjective Surgeon Satisfaction will be rated from 0 to 10. (0= not satisfied, 10= very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Berit Schneider-Stickler, Dr., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No